CLINICAL TRIAL: NCT00748046
Title: Phase 1, Open-label, Single Ascending-dose Study to Assess Safety, Pharmacokinetics, Biodistribution and Radiation Dosimetry of Intravenous Doses of Alpharadin™ Injection (Radium-223 Chloride) in Patients With HRPC and Skeletal Metastases
Brief Title: Alpharadin™ (Radium-223 Chloride) Safety and Dosimetry With HRPC That Has Metastasized to the Skeleton
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15303; BC1-08 (Other: Algeta ASA)
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Prostate Cancer; Metastases; Pharmacokinetics
Keywords: Biodistribution; Radiation dosimetry; Pharmacokinetics; Safety
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radium-223 chloride (Xofigo, BAY88-8223) (Experimental): The patients will receive Radium-223 chloride as an escalating dose of either 50, 100 or 200 kBq/kg b.w. (0.0014, 0.0027 or 0.0054 mCi/kg).
  Interventions: Drug: Radium-223 chloride (BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 chloride (BAY88-8223) — The required volume of study drug to be administered to a patient was calculated using the patient's body weight.

SUMMARY:
The purpose of the study is to investigate the safety, biodistribution, radiation dosimetry and pharmacokinetics of three intravenous escalating dose levels of Xofigo (Alpharadin).

DETAILED DESCRIPTION:
Within the U.S., the trial is conducted under an IND sponsored by Bayer.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥18 years of age
* Have histologically or cytologically evidence of adenocarcinoma of the prostate
* Have progressive castrate metastatic disease as shown by at least one of the following:

  * Imaging modalities:

    * Radionuclide Bone Scan: New osseous lesions
    * MRI or CT: At least a 20% increase in the sum of the LD of target lesions OR
  * Biochemical progression: A minimum of three rising PSA values from a baseline that are obtained 1 week or more apart, or 2 measurements 2 or more weeks apart
* Have skeletal metastases confirmed by bone scintigraphy within the last 4 weeks. Evidence of at least 2 bone metastases on bone scan.
* Have castrate levels of testosterone (<50 ng/ml). Treatment to maintain castrate levels of testosterone must be continued.
* Patients who have failed initial hormonal therapy using either an orchiectomy or a GnRH agonist in combination with an antiandrogen must first progress through antiandrogen withdrawal prior to being eligible. The minimum timeframe to document failure of anti-androgen withdrawal will be four weeks.
* Have Karnofsky performance status ≥60%
* Have a life expectancy ≥6 months
* Have the following laboratory requirements:

  * White Blood Count (WBC) ≥3,000/mm3
  * Absolute Neutrophil Count (ANC) ≥1,500/ mm3
  * Platelet (PLT) ≥100,000/ mm3
  * Hemoglobin (HGB) ≥10 mg/dl
  * Bilirubin ≤2.0 mg/dl (unless the patient has Gilbert's syndrome)
  * AST and ALT ≤2,5 times upper institutional limit of the normal range
  * Serum creatinine ≤2.0 mg/dl
* Must be able and willing to sign an informed consent indicating that he is aware of the investigational nature of this study in keeping with the policies of the institution and have provided written authorization for use and disclosure of protected health information
* Must be willing and able to comply with the protocol, and agrees to return to the hospital for follow-up visits and examination

Exclusion Criteria:

* Have received an investigational drug within 4 weeks prior to the administration of Radium-223 chloride, or is scheduled to receive one during the treatment and post-treatment period
* Have received chemo-, immunotherapy, or external radiotherapy within the last 4 weeks prior to administration of study drug, or has not recovered from acute adverse events as a result of such therapy
* Have received prior hemibody external radiotherapy
* Have a need for immediate external radiotherapy
* Have received systemic radiotherapy with radium-223, strontium-89, samarium-153, rhenium-186 or rhenium-188 for the treatment of bony metastases within the last 24 weeks prior to administration of study drug
* When receiving bisphosphonates, have changed the dose within 4 weeks before administration of study drug
* Have started or stopped systemic steroids within a week prior to study drug administration, or are expected to be subject to changes in the systemic steroid medication
* Have imminent or established spinal cord compression based on clinical findings and/or MRI
* Have other currently active (relapse within the last 3 years) malignancy (except non-melanoma skin cancer) that are not prostate cancer metastases
* Have small cell carcinoma
* Have predominant visceral metastases (≥ 3 lung or liver lesions) or symptomatic lymph-adenopathy (scrotal or pedal edema)
* Any other serious illness or medical condition, for example:

  * any uncontrolled infection
  * any patient who has clinical heart failure severe enough to cause marked limitation of activity, and who is only comfortable at rest; or any patient who has heart failure more severe than this (NYHA Heart Failure Class III or IV)
  * Crohn's disease or ulcerative colitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
All safety data, including adverse events, occurrence of treatment-emergent adverse events, changes in laboratory variables, vital signs, ECG, physical examination, long term radiation toxicity, including results of bone marrow biopsy | 1 year
Biodistribution, dosimetry and pharmacokinetics (whole body activity assessment, the counts in region-of-interest (ROIs) from anterior and posterior whole-body images, and the assay of activity in blood | 6 days after injection

SECONDARY OUTCOMES:
Post-treatment PSA effect: PSA decline, time to PSA progression after PSA response | 1 year
Post-treatment bone markers effect: Changes in bone marker values from pre- to post administration | 1 year
Circulating tumor cells (CTCs) enumeration and role of molecular profiling of CTC in predicting sensitivity to treatment and treatment response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Morris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- New York, New York, United States

REFERENCES:
- [Result] Carrasquillo JA, O'Donoghue JA, Pandit-Taskar N, Humm JL, Rathkopf DE, Slovin SF, Williamson MJ, Lacuna K, Aksnes AK, Larson SM, Scher HI, Morris MJ. Phase I pharmacokinetic and biodistribution study with escalating doses of (2)(2)(3)Ra-dichloride in men with castration-resistant metastatic prostate cancer. Eur J Nucl Med Mol Imaging. 2013 Sep;40(9):1384-93. doi: 10.1007/s00259-013-2427-6. Epub 2013 May 8. PMID 23653243